CLINICAL TRIAL: NCT02251496
Title: Oral Nutrition Supplements vs. Energy- and Protein Dense in Between Meal Snacks, Weight Changes and Functional Capacity in Chronic Obstructive Pulmonary Disease; Randomized Controlled Dietary Intervention
Brief Title: COPD: Oral Nutrition Supplements vs. Energy- and Protein Dense in Between Meal Snacks.
Acronym: COPD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Iceland (Other)
Responsible Party: Principal Investigator, Áróra Rós Ingadóttir, Nutritionist M.Sc, University of Iceland
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: COPD-141316051
Record Dates: First submitted 2014-09-25; First posted 2014-09-29 (Estimated); Results first posted 2021-01-19 (Actual); Last update posted 2021-01-19 (Actual); Status verified 2020-12

CONDITIONS: Malnutrition
Keywords: Malnutrition; Chronic obstructive pulmonary disease; Nutrition Therapy; Oral Nutrition Supplement; Food
MeSH Terms: conditions — Malnutrition; Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Oral nutrition supplement (ONS-group) (Active Comparator): The subjects in this group will be provided with and encouraged to take two ready to drink oral nutrition supplements (ONS) daily, providing ~ 600 kcal/d in addition to the hospital food (during hospitalisation) or in addition to their daily diet at home (after discharge from the hospital).
  Interventions: Other: Oral nutrition supplement (ONS-group)
- In between meals snacks (Snacks-group) (Active Comparator): In between meals snacks (Snacks-group): The subjects in this group will be provided with and encouraged to select in-between-meals snacks providing ~ 600 kcal/d in addition to the hospital food (during hospitalisation) or in addition to their daily diet at home (after discharge from the hospital).
  Interventions: Other: In between meals snacks (Snacks-group)

INTERVENTIONS:
Other: In between meals snacks (Snacks-group) — In between meals snacks (Snacks-group): The subjects in this group will be provided with and encouraged to select in-between-meals snacks providing ~ 600 kcal/d in addition to the hospital food (during hospitalisation) or in addition to their daily diet at home (after discharge from the hospital).
  Arms: In between meals snacks (Snacks-group)
Other: Oral nutrition supplement (ONS-group) — The subjects in this group will be provided with and encouraged to take two ready to drink oral nutrition supplements (ONS) daily, providing ~ 600 kcal/d in addition to the hospital food (during hospitalisation) or in addition to their daily diet at home (after discharge from the hospital).
  Arms: Oral nutrition supplement (ONS-group)

SUMMARY:
At least one fifth of patients in European hospitals are malnourished. Malnutrition is associated with negative consequences, including higher rates of complications, longer hospital stay, impaired wound healing and increased mortality with consequent effects on costs of healthcare. Evidence suggests that there may be benefits to some malnourished patients from receiving oral nutrition supplements in the short-term but it is not known whether these benefits can be sustained and indeed whether similar benefits may be achieved using food-based interventions of lower cost. The overall objective of the study is to compare two nutritional interventions among malnourished patients with COPD (n=200); oral nutrition supplement (ONS) vs. energy and protein dense in-between meals snack during hospitalisation and at home. Subjects will be followed for one year. The primary endpoint is weight change. Secondary endpoints include forced expiratory volume in one second, forced vital capacity, six-minute walk distance, hand-grip strength, health related quality of life, length of hospital stay, energy- and protein intake, readmissions to the hospital and acute exacerbation. No studies are available comparing the supply of ONS to malnourished patients with COPD compared with the provision of regular food (in-between meals snacks). The results of the study will provide important information that might improve nutrition care in the hospital setting as well as after discharge from the hospital

DETAILED DESCRIPTION:
Patients with established COPD admitted to the Department of Pulmonary Medicine at Landspitali National University Hospital from September 2014-September 2016 will be screened for malnutrition using the NRS2002 screening tool, recommended by ESPEN. Those identified at risk of malnutrition and are able to give informed consent will be recruited. According to the Hospital statistics and previous studies on the frequency of malnutrition in this patient group, the time frame for recruitment is long enough to recruit 200 subjects who will be randomised into the two study groups (~ 3 subjects per week).

The following baseline data will be collected in order to identify possible confounders. This will include; socio-demographic data (age, gender, civil status, household size, family and social network); major medical diagnosis; use of medication; GOLD score (Global Initiative for Chronic Obstructive Lung Disease), depressive symptoms, cognition), additional discharge interventions (e.g. outgoing hospital teams, day care with exercise); and use of oral nutritional supplements.

Inclusion criteria are:

* Newly admitted patients > 18 years old who were at nutritional risk according to the validated nutritional risk screening tool (NRS-2002, score 3+)
* Able to eat orally
* An anticipated length of hospitalization of > 3 days
* Sufficient language proficiency

Exclusion criteria are:

* Dysphagia
* Food allergy or intolerance
* Anatomical obstructions preventing oral food intake Exclusion during follow-up: Subjects who withdraw their consent to participate.

Outcome measures:

The primary endpoint is weight changes up to one year from admission to the hospital. Secondary endpoints include forced expiratory volume in one second (FEV1), forced vital capacity (FVC), six-minute walk distance, hand-grip strength, health related quality of life (HRQoL), length of hospital stay, nutritional status, energy- and protein intake, readmissions to the hospital in within 30 days, as well as the total number of readmissions to the hospital and acute exacerbation during follow-up. Functional outcome measurements will be conducted by trained research assistant in collaboration with the PhD student. Information about background diets, HRQoL as well as compliance to the intervention diets will be gathered by the PhD and MS students.

Measurements will be conducted at admission to the hospital (baseline measurements) and before discharge from the hospital. Clinical examinations at Landspitali National University Hospital are planned 3, 6 and 12 months after discharge from the hospital. All together we aim at having five measurement points for each subject. Each examination will take ~ 80 minutes (30 min for the FEV1 and FVC tests, 20 min for the walking test and measurement of hand-grip strength, and 30 min for the 24-hour recalls and HRQoL questionnaires). Additionally, the subjects will be contacted on at least two other occasions by phone, in weeks 2 and 6 (each interview ~20 min).

ELIGIBILITY:
Inclusion Criteria:

* Newly admitted patients > 18 years old who were at nutritional risk according to the validated nutritional risk screening tool (NRS-2002, score 3+)
* Able to eat orally
* An anticipated length of hospitalization of > 3 days
* Sufficient language proficiency

Exclusion Criteria:

* Dysphagia
* Food allergy or intolerance
* Anatomical obstructions preventing oral food intake

Exclusion during follow-up: Subjects who withdraw their consent to participate.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2014-09; Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Áróra R Ingadóttir, Master, Principal Investigator — Unit for Nutrition Research (UNR)
Locations (1):
- The Department of Thoracic Medicine at Landspítali, Reykjavik, Iceland

REFERENCES:
- [Result] Ingadottir AR, Beck AM, Baldwin C, Weekes CE, Geirsdottir OG, Ramel A, Gislason T, Gunnarsdottir I. Oral nutrition supplements and between-meal snacks for nutrition therapy in patients with COPD identified as at nutritional risk: a randomised feasibility trial. BMJ Open Respir Res. 2019 Jan 3;6(1):e000349. doi: 10.1136/bmjresp-2018-000349. eCollection 2019. PMID 30687503

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Oral Nutrition Supplement (ONS-group) | In Between Meals Snacks (Snacks-group)
Started | 19 | 15
Completed | 14 | 11
Not Completed | 5 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Oral Nutrition Supplement (ONS-group) | In Between Meals Snacks (Snacks-group) | Total
Number analyzed (Participants) | 19 | 15 | 34
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 19 | 15 | 34
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 11 | 24
  Male | 6 | 4 | 10
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Iceland | 19 | 15 | 34
Weight [Mean (Standard Deviation); unit: kg] | 54 (10) | 49 (10) | 51.4 (9.9)
BMI [Mean (Standard Deviation); unit: kg/m^2] | 19.4 (4.1) | 18.0 (2.7) | 18.8 (3.5)

OUTCOME MEASURES:

1. Primary Outcome: Weight Changes
Description: Weight changes from baseline and one year from admission to the hospital
Time Frame: baseline and one year from admission to the hospital
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Oral Nutrition Supplement (ONS-group) | In Between Meals Snacks (Snacks-group)
Number analyzed (Participants) | 19 | 15
kg | 2.3 (4.6) | 4.4 (6.4)

2. Secondary Outcome: Health Related Quality of Life (HRQoL)
Description: Saint George's Respiratory Questionnaire total score (SGRQ) This validated questionnaire is based on 76 items used to calculate three component scores: symptoms, activity and impact, and a total score. A score of 100 represents worst possible health status and a score of 0 represents best possible health status. A change of 4 points in the SGRQ total score is considered the minimum clinically relevant difference.
Time Frame: baseline and one year from admission to the hospital
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Oral Nutrition Supplement (ONS-group) | In Between Meals Snacks (Snacks-group)
Number analyzed (Participants) | 19 | 15
score on a scale | 3.9 (11.1) | 8.9 (14.1)

ADVERSE EVENTS:
Time Frame: 12 months
Description: The number of participants at risk for Serious Adverse Events and at risk for Other (Not Including Serious) Adverse Events is 34.
Arm/Group | Oral Nutrition Supplement (ONS-group) | In Between Meals Snacks (Snacks-group)
All-Cause Mortality (participants affected / at risk) | 4/19 | 3/15
Serious Adverse Events (participants affected / at risk) | 0/19 | 0/15
Other Adverse Events (participants affected / at risk) | 0/19 | 0/15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2020-12-23): https://cdn.clinicaltrials.gov/large-docs/96/NCT02251496/Prot_000.pdf
  • Statistical Analysis Plan (2020-12-23): https://cdn.clinicaltrials.gov/large-docs/96/NCT02251496/SAP_001.pdf